CLINICAL TRIAL: NCT00457717
Title: Myopia Control by Combining Auricular Acupoint and Atropine Eyedrops
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMR94-IRB-49
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Myopia
Keywords: myopia, auricular acupoint, atropine, RCT
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 0.25 % atropine
Drug: 0.5 % atropine
Procedure: 0.25 % atropine+auricular acupoints

SUMMARY:
This study was designed to compare the difference of using atropine eyedrops alone from atropine combined with the stimulation of auricular acupoints therapy in reducing myopia progression.

DETAILED DESCRIPTION:
A total of 64 school-aged children with myopia, fulfilling eligibility criteria, were recruited. They were randomly assigned to three arms:

1. 21 treated with the 0.25 % atropine each night (0.25A).
2. 20 treated with the 0.5 % atropine each night (0.5A).
3. 23 treated with 0.25 % atropine each night together with stimulation of auricular acupoints(0.25A+E).

This protocol was proceeded for at least 6 months.The differences in post-treatment effects of these three groups were statistically accessed.

ELIGIBILITY:
Inclusion Criteria:

* all included patients, age from 6 to 15 years, had myopia (spherical equivalent > -0.5 D) after cycloplegic refraction,
* The astigmatism and anisometropia were less than 2.0 D,
* IOP was less than 21 mmHg.

Exclusion Criteria:

* the presence of related disease such as infection, ulceration, eyelid disease, ocular and auricular disorders,
* individuals with amblyopia or strabismus,
* individuals received any other therapies in the period of study,
* individuals suffering some sort of haemostasis disorder,
* individuals did not follow the treatment (eyedrops and/or stimulation of auricular acupoints) over seven days

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2005-07; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
the progression of myopia degree, axial length elongation of eye

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Liang Chang, PhD, Principal Investigator — China Medical University, Taiwan
Locations (1):
- China Medical University, Taichung, Taiwan

REFERENCES:
- [Background] Goss DA. Attempts to reduce the rate of increase of myopia in young people--a critical literature review. Am J Optom Physiol Opt. 1982 Oct;59(10):828-41. doi: 10.1097/00006324-198210000-00010. PMID 7148977
- [Background] Lin LL, Shih YF, Hsiao CK, Chen CJ. Prevalence of myopia in Taiwanese schoolchildren: 1983 to 2000. Ann Acad Med Singap. 2004 Jan;33(1):27-33. PMID 15008558
- [Background] Saw SM, Shih-Yen EC, Koh A, Tan D. Interventions to retard myopia progression in children: an evidence-based update. Ophthalmology. 2002 Mar;109(3):415-21; discussion 422-4; quiz 425-6, 443. doi: 10.1016/s0161-6420(01)00972-1. PMID 11874738
- [Result] Shih YF, Chen CH, Chou AC, Ho TC, Lin LL, Hung PT. Effects of different concentrations of atropine on controlling myopia in myopic children. J Ocul Pharmacol Ther. 1999 Feb;15(1):85-90. doi: 10.1089/jop.1999.15.85. PMID 10048351
- [Result] Chen MC. 112 cases of juvenile myopia treated by auricular acupressure. J Tradit Chin Med. 1989 Sep;9(3):173. No abstract available. PMID 2615447
- [Derived] Liang CK, Ho TY, Li TC, Hsu WM, Li TM, Lee YC, Ho WJ, Cheng JT, Tzeng CY, Liu IT, Chang SL. A combined therapy using stimulating auricular acupoints enhances lower-level atropine eyedrops when used for myopia control in school-aged children evaluated by a pilot randomized controlled clinical trial. Complement Ther Med. 2008 Dec;16(6):305-10. doi: 10.1016/j.ctim.2008.04.007. Epub 2008 May 29. PMID 19028329